



This model informed consent form has been reviewed by the DCT/NCI and is the official consent document for this study. Institutions must use the sections of this document that are in bold type in their entirety. Editorial changes to these sections may be made as long as they do not change information or intent. If the local IRB insists on making deletions or more substantive modifications to any of the sections in bold type, they must be justified in writing by the investigator at the time of the institutional audit.

#### SAMPLE RESEARCH INFORMED CONSENT/PARENTAL PERMISSION FORM

PEPN1812, A Phase 1 Trial of the CD123 X CD3 DART® Molecule Flotetuzumab (NSC#808294, page 125) in Children, Adolescents, and Young Adults with Relapsed or Refractory Acute Myeloid Leukemia

If you are a parent or legal guardian of a child who may take part in this study, permission from you is required. The assent (agreement) of your child may also be required. When we say "you" in this consent form, we mean you or your child; "we" means the doctors and other staff.

## Overview

You are being asked to take part in this research study because you have been diagnosed with leukemia that has either come back ("relapsed") or does not respond to therapy (is "refractory").

Taking part in this study is voluntary. You may choose not to be in this study. If you decide not to be in this study, you will not be penalized and you will not lose any benefits to which you are entitled. You will still receive medical care.

The overall goal of this study is to find the highest dose of the experimental drug, flotetuzumab, that we can give safely. This study is called a Phase 1 study. A description of the goals of a Phase 1 study can be found in the section Why is this study being done? Flotetuzumab has not been approved for use by the FDA for adults or for children. If there is no improvement in your leukemia after 2 cycles of treatment, your treatment with flotetuzumab will be stopped.

If the exams, tests and procedures show that you can be in the study, and you choose to take part, flotetuzumab will be given by vein continuously for 28 days, with the infusion ending on Day 29. This entire 29 day period is called a cycle. After infusion ends on Day 29 you will receive a treatment-free period for up to 3 days. Your doctor will decide exactly how many days you will go without taking flotetuzumab but it will be no more than 3 days. Alternatively, your doctor may decide that it is in your best interest to have no treatment-free days. You may continue to receive flotetuzumab for up to 6 cycles (with your doctor determining the length of your treatment-free period at the end of each cycle) unless you develop serious side effects or your cancer worsens.





Before you begin the first cycle you will also be given the commercial drug, cytarabine, into the spinal fluid. Your doctor will decide if you should keep receiving cytarabine before each subsequent cycle.

The dose for the first children enrolled on the study will be based on the side effects seen in adults. We will be looking at up to 3 different dose levels of flotetuzumab, depending on the side effects we see in the children on this study. Between 2 and 6 children will receive flotetuzumab at each dose. If the side effects are not too severe, the next group of children will receive a higher dose. Dosing is done this way because we do not yet know the best dose to use in children.

If you are enrolled early in this study you may receive a lower dose than those who are enrolled later. A lower dose may be less likely to have any effect on your cancer. If you are enrolled in this study at a high dose level you may be more likely to have side effects. If you have bad side effects, your dose may be decreased. Up to 3 different doses of flotetuzumab may be studied. During the 7-8 days of the first cycle, there will be a slow increase in the medication to your goal dose, but outside of this time period, there will be no increases in the medication.

All people who receive cancer treatment are at risk of having side effects. In addition to killing tumor cells, cancer chemotherapy can damage normal tissue and produce side effects.

This study uses the investigational drug, flotetuzumab. One common side effect of this drug is that patients experience a reaction following infusion of the drug that causes fever, chills, rash, or low blood pressure. Other common side effects are fever and nausea. A less common but serious side effect is something called "cytokine release syndrome" which is characterized by fevers and may include low blood pressure and/or low oxygen levels. The full list of risks for flotetuzumab are available in the section What side effects or risks can I expect from being in the study?

You can ask your study doctor questions about side effects at any time.

We hope that this study will help you personally, but we do not know if it will. The potential benefits to you associated with participation in this study are described in the section <u>Are there benefits to taking part in the study?</u>

You have a choice between another treatment for leukemia and this clinical trial.

The rest of this form provides detailed information about the study and what to expect should you decide to participate.

# Why am I being invited to take part in this study?

You are being asked to take part in this research study because you have been diagnosed with leukemia that has either come back ("relapsed") or does not respond to therapy (is "refractory").

This study is called a clinical trial. A clinical trial is a research study involving treatment of a disease in human patients. This study is being carried out by the Children's Oncology Group (COG) Pediatric Early Phase Clinical Trial Network (PEP-CTN). COG is an international research group that consists of more than 200 hospitals that treat children with cancer in the United States, Canada, Australia, and Switzerland. The PEP-CTN is the group within COG that





consists of 21 hospitals based in the United States and Canada, and participation in this study will be limited to these hospitals.

It is common to enroll children and adolescents with cancer in a clinical trial that seeks to improve cancer treatment over time. Clinical trials include only people who choose to take part. You have a choice between another treatment for leukemia and this clinical trial.

Please take your time to make your decision. You may want to discuss it with your friends and family. We encourage parents to include their child in the discussion and decision to the extent that the child is able to understand and take part.

## What is the current standard of treatment for this disease?

We are asking if you want to participate in this study because there is not a standard treatment for your cancer at this point.

# Why is this study being done?

This is a Phase 1 study of a drug called flotetuzumab. We are testing new experimental drugs such as flotetuzumab in the hopes of finding a treatment that may be effective against leukemia that has come back or that has not responded to standard therapy. This study looks at how well flotetuzumab works when given to children and young adults with relapsed or refractory leukemia. Flotetuzumab is experimental because it has not been proven to work in a situation like yours. We are using flotetuzumab because it seems to work against cancer in test tubes and animals. Flotetuzumab has been used in adults and there is a lot that we do not know about it yet. This is called a Phase 1 study because the goal is to find the highest dose of flotetuzumab that we can give safely.

## The overall goals of this study are to

- Find the highest safe dose of flotetuzumab that can be given without causing severe side effects;
- Learn what kind of side effects flotetuzumab can cause;
- Learn more about the pharmacology (how your body handles the drug) of flotetuzumab;
- Learn more about the effects of flotetuzumab on your immune system;
- Determine whether flotetuzumab is a beneficial treatment for your cancer

# What will happen on this study that is research?

If the exams, tests and procedures show that you can be in the study, and you choose to take part, flotetuzumab will be given by vein/central line continuously for 28 days, with the infusion ending on Day 29. This entire 29 day period is called a cycle. After infusion ends on Day 29 you will receive a treatment-free period for up to 3 days. Your doctor will decide exactly how many days you will go without taking flotetuzumab but it will be no more than 3 days. Alternatively, your doctor may decide that it is in your best interest to have no treatment-free days. You may





continue to receive flotetuzumab for up to 6 cycles (with your doctor determining the length of your treatment-free period at the end of each cycle) unless you develop serious side effects or your cancer worsens.

Before you begin the first cycle you will also be given the commercial drug, cytarabine, into the spinal fluid. Your doctor will decide if you should keep receiving cytarabine before each subsequent cycle.

You will need a special kind of IV called a "central line." This is a special kind of IV placed into a big vein in your chest that can stay in for a long time. If you get a central line, you will have a separate consent form for it.

You will need to remain in the hospital for the entirety of Cycle 1. For subsequent cycles, your doctor will decide if you can receive your flotetuzumab treatments at home. Even if you are able to receive your flotetuzumab treatments at home for subsequent cycles, you will still need to return to the hospital every 96 hours to have your flotetuzumab infusion bag changed.

## **Dose Escalation/ Dose Confirmation**

The dose for the first children enrolled on the study will be based on the side effects seen in adults. We will be looking at up to 3 different dose levels of flotetuzumab, depending on the side effects we see in the children on this study. Between 2 and 6 children will receive flotetuzumab at each dose. If the side effects are not too severe, the next group of children will receive a higher dose. Dosing is done this way because we do not yet know the best dose to use in children. If you are enrolled early in this study you may receive a lower dose than those who are enrolled later. A lower dose may be less likely to have any effect on your cancer. If you are enrolled in this study at a high dose level you may be more likely to have side effects. If you have bad side effects, your dose may be decreased. Up to 3 different doses of flotetuzumab may be studied. Future patients will be treated at the highest dose level that is deemed tolerable to patients on this study. During the first 7 – 8 days of the first cycle, there will be a slow increase in the medication to your goal dose, but outside of this time period, there will be no planned increases in the medication. If your doctor chooses to extend your treatment-free period between cycles by more than 3 days, the slow increase in the medication to your goal dose will be done again for the first cycle after your extended treatment-free period.





## **Diagram of Treatment**

An overview of a treatment cycle is below:

## The table below describes one cycle of therapy:

| Drug | How the drug will be given | Days |
|---|---|---|
| Cytarabine | Into the spinal fluid (intrathecal) | Prior to flotetuzumab therapy for Cycle 1* |
| Flotetuzumab | By vein/central line | 1-29 |

<sup>\*</sup>Your doctor will decide if you should receive cytarabine prior to subsequent cycles.

## **Research Study Tests and Procedures**

During the study you will have tests and procedures to check for side effects and see how your cancer is doing. These tests are part of regular cancer care, but you may have them more often because you are on the study:

- Physical exam
- Vital signs (blood pressure, pulse, temperature)
- Blood tests
- Pregnancy test (for females of child bearing age)
- MRI, X-rays, CT scans, or other tests that are needed to check your leukemia
- Bone marrow tests
- Heart function test (ECHO and EKG)
- Neurologic exam

Copies of the scans used to diagnose your cancer and some of the tissue already taken may be sent to a central review center. COG PEP-CTN does this to double check the hospitals' results and they are for research purposes only.



<sup>\*</sup>Required prior to Cycle 1 only. You may receive your dose of intrathecal cytarabine up to 1 week prior to starting flotetuzumab treatment. Additional doses of intrathecal cytarabine are optional during subsequent cycles. Your doctor will decide if you should receive cytarabine prior to subsequent cycles.

<sup>^</sup>Your doctor will decide exactly how many days you will go without taking flotetuzumab. Alternatively, your doctor may decide that you do not need any treatment-free days.





# **Required Research Study Tests**

The following tests will be done because you are part of this study. If you were not in the study you would probably not have these tests. The information learned would not change the way you are treated, and the results of these tests will not be given to you. You and your insurance company will not be charged for the costs of the required research study tests listed below.

#### **Pharmacokinetic Studies**

During this study we will use some of your blood to do tests called pharmacokinetic tests. Pharmacokinetic tests determine how much of the flotetuzumab is in your blood. Pharmacokinetic blood samples will be required from all participants in the study. Because we cannot draw the samples from the central line we give the drug through, we will start a separate IV to get the samples. Depending on what dose of flotetuzumab you are receiving, you will be put on 1 of 3 different pharmacokinetic testing schedules. Your study doctor will let you know which schedule you will follow. The 3 schedules are listed below:

<u>Pharmacokinetic Schedule #1</u>: Blood samples (about 2-3 mL or about  $\frac{1}{2}$  teaspoon each sample) will be collected before infusion begins on Cycle 1 Day 1, and on Days 3-8, 12, 15, 19, 22, 27, and 29 of Cycle 1. Blood samples will also be taken 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours after the end of infusion on the last day of your last cycle of therapy.

Depending on how long you are in the study, if you are on Pharmacokinetic Schedule #1, a total volume of 26 - 57 mL (about  $5 - 11\frac{1}{2}$  teaspoons) will be drawn for pharmacokinetic tests in this study. This amount of blood is safe to draw even from small children.

<u>Pharmacokinetic Schedule #2:</u> Blood samples (about 2-3 mL or about  $\frac{1}{2}$  teaspoon each sample) will be collected before infusion begins on Cycle 1 Day 1, and on Days 4, 6, 8, 9, 13, 17, 21, 25, and 29 of Cycle 1. Blood samples will also be taken 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours after the end of infusion on the last day of your last cycle of therapy.

Depending on how long you are in the study, if you are on Pharmacokinetic Schedule #2, a total volume of 20 – 48 mL (about 4 – 10 teaspoons) will be drawn for pharmacokinetic tests in this study. This amount of blood is safe to draw even from small children.

<u>Pharmacokinetic Schedule #3:</u> Blood samples (about 2-3 mL or about  $\frac{1}{2}$  teaspoon each sample) will be collected before infusion begins on Cycle 1 Day 1, and on Days 3-9, 13, 17, 21, 25, and 29. Blood samples will also be taken 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, and 24 hours after the end of infusion on the last day of your last cycle of therapy.

Depending on how long you are in the study, if you are on Pharmacokinetic Schedule #3, a total volume of 26 - 57 mL (about  $5 - 11\frac{1}{2}$  teaspoons) will be drawn for pharmacokinetic tests in this study. This amount of blood is safe to draw even from small children.





## **Immunogenicity Studies**

During this study we will use some of your blood to do tests called immunogenicity tests. Immunogenicity tests determine how your immune system reacts to flotetuzumab. Immunogenicity blood samples will be required from all participants in the study. Because we cannot draw the samples from the same IV or central line we give the drug through, we will start a separate IV to get the samples. Blood samples (2 - 3 mL) or about  $\frac{1}{2}$  teaspoon each sample) will be collected before infusion begins on Day 1 of Cycles 1, 3, and 5.

A total blood volume of 6 - 9 mL (about 1 - 2 teaspoons) will be drawn for immunogenicity tests in this study. This amount of blood is safe to draw even from small children.

## **Optional Research Study Tests**

We would also like to do some tests called biologic tests. These tests are important to help us learn more about flotetuzumab and may help children and young adults who receive flotetuzumab in the future. The information learned would not change the way you are treated, and the results of these tests will not be given to you. You do not have to do these tests if you do not want to. You can still be in the study if you do not want to do these tests. At the end of this consent form, there is a place to record your decision about taking part in each test. You and your insurance company will not be charged for the costs of the optional research study tests listed below.

During the study we would like to collect additional blood and bone marrow samples to evaluate the effect of flotetuzumab on your body. There are 5 different studies we would like your blood or bone marrow samples for, and you can participate in any, all, or none of the studies.

#### **Residual Leukemia Identification Study**

The first study will help us identify any residual leukemia by genetic testing after treatment with flotetuzumab, even if it is at very low levels. The bone marrow samples, 10 - 15 mL each (about 2 - 3 teaspoons), will be obtained prior to Cycle 1 and at the end of each cycle at the time of bone marrow evaluation.

A total bone marrow volume of 70-105 mL (about 14-21 teaspoons) will be drawn for this residual leukemia identification study. This amount of bone marrow is safe to draw even from small children. If bone marrow cannot be obtained prior to Cycle 1, your doctor may draw blood instead for this time point only. If this is the case, you will have 20-30 mL (about 4-6 teaspoons) of blood drawn prior to Cycle 1 and 60-90 mL (about 12-18 teaspoons) of bone marrow drawn throughout the rest of the study for these residual leukemia tests. This amount of bone marrow and blood is safe to draw even from small children.

This study will include research about genes. Genes carry information about features that are found in you and in people who are related to you. Some of your genetic and health information may be placed in central databases that may be made available to qualified researchers, along with information from many other people. Information that could directly identify you will not be included.

Even without your name or other identifiers, your genetic information is unique to you. If you agree to Biobanking, there is a risk of a data security breach and that someone could trace the genetic information in a central database back to you. Although this has never happened in real





8

life and we have many safeguards in place to prevent it from happening, the risk may change in the future as people come up with new ways of tracing information. There are laws against the misuse of genetic information, but they may not give full protection. In some cases, misuse of the information could be used to make it harder for you to get or keep a job or insurance.

There can also be risks in learning about your own genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a study. Sometimes this is upsetting to families or they wish they didn't know the information. We encourage you to discuss this study with your relatives before you decide whether to participate in the Biobanking part.

If you want to learn more about tissue research with banked specimens, the NCI website has an information sheet called "Providing Your Tissue For Research: What You Need To Know." This sheet can be found at: <a href="http://www.cancer.gov/clinicaltrials/resources/providingtissue">http://www.cancer.gov/clinicaltrials/resources/providingtissue</a>.

## Leukemia: Immune Cell Ratio Study

The second study will help us determine the ratio of leukemia cells you have in comparison to certain immune cells. The blood samples, 2-3 mL each (about  $\frac{1}{2}$  teaspoon), will be obtained prior to flotetuzumab treatment on Day 1 of each cycle, and on Days 8, 14, 22, and 29 of Cycle 1.

A total volume of 28 – 42 mL (about 6 - 9 teaspoons) will be drawn for this leukemia:immune cell ratio study. *This amount of blood is safe to draw even from small children*.

#### **Immune System Study**

The third study will help us evaluate how your immune system responds to flotetuzumab by measuring the proteins that are secreted by your immune cells. The blood samples will be obtained prior to flotetuzumab treatment on Cycle 1 Day 1, and on Cycle 1 Day 8. The blood samples will total 2-3 mL each (about ½ teaspoon). Additionally, if you experience an infusion-related reaction to flotetuzumab, we would also like to collect blood samples at the time of the reaction and when the reaction is resolved.

A total volume of 4 - 12 mL (about  $1 - 2\frac{1}{2}$  teaspoons) will be drawn for this immune system study. This amount of blood is safe to draw even from small children.

#### **Biological Marker Study**

The fourth study will help us figure out if there are any specific biological markers in your bone marrow prior to the start of therapy that would predict a response to flotetuzumab. The bone marrow samples will be obtained prior to Cycle 1 and will be used for further genetic testing and for the growing of your leukemia cells in mouse models in the research laboratory.

A total bone marrow volume of 10-15 mL (about 2-3 teaspoons) will be drawn for this biological marker study. This amount of bone marrow is safe to draw even from small children. If bone marrow cannot be obtained prior to Cycle 1, your doctor may draw blood instead. If this is the case, you will have a total of 20-30 mL (about 4-6 teaspoons) of blood drawn for this biological marker study. This amount of blood is safe to draw even from small children.





# Flotetuzumab Target Quantification Comparison Study

The fifth study will help us quantify how much of the flotetuzumab target (CD123) your leukemia is expressing prior to flotetuzumab therapy which we will associate with response to therapy. The bone marrow samples will be obtained prior to Cycle 1.

A total bone marrow volume of 5 mL (about 1 teaspoon) will be drawn for this flotetuzumab target quantification comparison study. *This amount of bone marrow is safe to draw even from small children.* If bone marrow cannot be obtained prior to Cycle 1, your doctor may draw blood instead. If this is the case, you will have 10 mL (about 2 teaspoons) of blood drawn for this flotetuzumab target quantification comparison study. *This amount of blood is safe to draw even from small children.* 

The table below summarizes the blood volume and bone marrow volume required if you participate in all of the above studies:

| Research Study | Preferred<br>Sample Type | Volume per<br>Sample | Total Volume |
|---|---|---|---|
| Pharmacokinetics | Blood | 2 – 3 mL | 20 – 57 mL |
| Immunogenicity | Blood | 2 – 3 mL | 6 – 9 mL |
| Residual Leukemia<br>Identification | Bone Marrow | 10 – 15 mL | 70 – 105 mL |
| Leukemia: Immune Cell<br>Ratio | Blood | 2 – 3 mL | 28 – 42 mL |
| Immune System | Blood | 2 – 3 mL | 4 – 12 mL |
| Biological Marker | Bone Marrow | 10 – 15 mL | 10 – 15 mL |
| Flotetuzumab Target<br>Quantification<br>Comparison | Bone Marrow | 5 mL | 5 mL |
| Total Volume for All<br>Studies | | | 143 – 245 mL |





# What side effects or risks can I expect from being in the study?

## **Treatment Risks**

All people who receive cancer treatment are at risk of having side effects. In addition to killing tumor cells, cancer treatment can damage normal tissue and produce side effects.

The most common serious side effect from cancer treatment is lowering of the number of blood cells resulting in anemia, increased chance of infection, and bleeding tendency. Low blood counts are described in the <a href="COG Family Handbook for Children with Cancer">COG Family Handbook for Children with Cancer</a>. Parents will be taught more about caring for their child when his or her blood counts are low.

## Risks of Study

You may lose time at school, work or home and spend more time in the hospital or doctor's office than usual. You may be asked sensitive or private questions which you normally do not discuss.

The cancer treatment used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drugs/study approach. Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

You can ask your study doctor questions about side effects at any time.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.
- The study doctor will provide you with information about other drugs you may need to avoid while receiving the study drugs.

The tables below show the most common and the most serious side effects that researchers know about in adults. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.













12

## Risks and side effects related to cytarabine when given into the spinal fluid (intrathecal):

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving cytarabine (ara-c) when given into the spinal fluid, more than 20 and up to 100 may have:

- Nausea, vomiting
- Fever
- Headache

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving cytarabine (ara-c) when given into the spinal fluid, from 4 to 20 may have:

- Anemia which may cause tiredness, or may require blood transfusions
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Tiredness, dizziness, loss of coordination
- Numbness and tingling of the arms and legs
- Inflammation of the lining of the brain that can lead to headache, numbness and tingling

#### RARE. AND SERIOUS

In 100 people receiving cytarabine (ara-c) when given into the spinal fluid, 3 or fewer may have:

- Seizure
- Paralysis
- Blurred vision with a chance of blindness
- Damage to the brain that may result in a decrease in the ability to learn

You must refrain from driving a motor vehicle or operating heavy machinery while receiving flotetuzumab treatment and for 30 days after your last dose of flotetuzumab.

In addition to the risks described above, there may be unknown risks, or risks that we did not anticipate, associated with being in this study.

#### Reproductive risks:

Women should not become pregnant and men should not father a baby while on this study because the drugs in this study can be bad for an unborn baby. If you or your partner can get pregnant, it is important for you to use birth control or not have sex while on this study and for 12 weeks after completion of flotetuzumab administration. Check with your study doctor about what kind of birth control methods to use. Some birth control methods might not be approved for use in this study. If you are a woman and become pregnant or suspect you are pregnant while participating in this study, please inform your treating physician immediately. Women should not breastfeed a baby while on this study. Also check with your doctor about how long you should not breastfeed after you stop the study treatment(s).





# Risks of blood drawing or placing an intravenous catheter for blood drawing: Risks associated with drawing blood are slight, but some risks include: pain, excessive bleeding, fainting or feeling lightheaded, bruising, infection (a slight risk any time the skin is broken), and multiple punctures to locate veins.

## **Bone Marrow Examination Risks:**

You will be required to take a bone marrow test for diagnostic purposes. You will be informed of the risks associated with the procedure and your study doctor will obtain a separate consent form.

### **Risks of Central Line Placement:**

Potential risks of central line placement include accumulation of air inside the chest; bleeding; infection; blood clot development in the line; and risks from the anesthesia. After placement, the central line may become infected which may require hospitalization, antibiotics and possibly removal and replacement of the central line.

For more information about risks and side effects, ask your study doctor.

# Are there benefits to taking part in the study?

We hope that this study will help you personally, but we do not know if it will.

Potential benefits to you could include:

- your cancer may stop growing or shrink for a period of time
- you may have lessened symptoms, such as pain, that are caused by the cancer

It is extremely unlikely that this treatment will cure your cancer. With any cancer treatment, sometimes treatment does not make the cancer go away. Or, sometimes treatment makes the cancer go away for a while but the cancer comes back later.

We expect that the information learned from this study will benefit other patients in the future.

# What other options are there?

Instead of being in this study, you have these options:

- Getting treatment for your cancer without being in a study.
- Taking part in another study.
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.





# How many people will take part in the study?

The total number of people enrolled on this study is expected to be between 4 and 47.

# How long is the study?

People in this clinical trial are expected to receive treatment on this study for about 6 months (6 cycles of therapy). After treatment, you will have follow-up examinations and medical tests.

We would like to continue to find out about your health for about 30 days after your last dose of flotetuzumab. By keeping in touch with you for a while after you complete treatment, we can better understand the long-term effects of the study treatments.

You can stop taking part in the study at any time. However, if you decide to stop participating in the study, we encourage you to talk to the study doctor and your regular doctor first. They will help you stop safely.

Your doctor or the study doctor may decide to take you off this study:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment
- if you experience side effects from the treatment that are considered too severe
- if new information becomes available that shows that another treatment would be better for you
- If your cancer gets worse
- If you become pregnant

# What about privacy?

We will do our best to make sure that the personal information in your medical record will be kept private. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. The Children's Oncology Group has a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the Children's Oncology Group will do their best to make sure that any information that goes out to others will not identify who you are. Information about this Certificate of Confidentiality is included in Attachment 1.

Organizations that may look at and/or copy your research or medical records for research, quality assurance and data analysis include groups such as:

- Children's Oncology Group and research partners
- The NCl's National Clinical Trials Network and the groups it works with to conduct research
- Representatives of the National Cancer Institute (NCI), Food and Drug Administration (FDA), and other U.S. and international governmental regulatory agencies involved in overseeing research.
- The Institutional Review Board of this hospital





- Pediatric Central Institutional Review Board (CIRB) of the National Cancer Institute
- The study sponsor and any drug company supporting the study or their designated reviewers.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

## What are the costs?

Taking part in this study may lead to added costs to you or your insurance company. There are no plans for the study to pay for medical treatment. Please ask about any expected added costs or insurance problems. Staff will be able to assist you with this.

In the case of injury or illness resulting from this study, emergency medical treatment is available but will be provided at the usual charge. No funds have been set aside to compensate you in the event of injury. However by signing this form, you are not giving up any legal rights to seek to obtain compensation for injury.

You or your insurance company will be charged for continuing medical care and/or hospitalization.

You will not be charged for the costs of the special blood studies and bone marrow studies that are being done for research purposes only, such as the pharmacokinetic and biology studies.

The drug company that makes flotetuzumab is supplying the drug at no charge for this study. The drug company does not cover the cost of getting the flotetuzumab ready and giving it to you, so you or your insurance company may have to pay for this.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at http://www.cancer.gov/clinicaltrials/learningabout.





# **Funding support**

If you choose to enroll on this study, this institution will receive some money from the PEP-CTN Children's Oncology Group to do the research. There are no plans to pay you for taking part in this study.

The drug company that makes flotetuzumab is providing money to the Children's Oncology Group to do the research.

This study includes providing specimens to the researcher, there are no plans for you to profit from any new product developed from research done on your specimens.

# What are my rights as a participant?

Taking part in this study is voluntary. You may choose not to be in this study. If you decide not to be in this study, you will not be penalized and you will not lose any benefits to which you are entitled. You will still receive medical care.

You can decide to stop being in the study at any time. Leaving the study will not result in any penalty or loss of benefits to which you are entitled. Your doctor will still take care of you.

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study. A committee outside of COG closely monitors study reports and notifies COG PEP-CTN if changes must be made to the study. Members of COG meet twice a year to discuss results of treatment and to plan new treatments.

# Whom do I call if I have questions or problems?

For questions about the study or if you have a research related problem or if you think you have been injured in this study, you may contact Dr. XXXX or your doctor at XXXX.

If you have any questions about your rights as a research participant or any problems that you feel you cannot discuss with the investigators, you may call XXXX Institutional Review Board (IRB) Administrator at XXXX.

If you have any questions or concerns that you feel you would like to discuss with someone who is not on the research team, you may also call the Patient Advocate at XXXX.

# Where can I get more information?

The <u>COG Family Handbook for Children with Cancer</u> has information about specific cancers, tests, treatment side effects and their management, adjusting to cancer, and resources. Your doctor can get you this Handbook, or you can get it at <a href="https://www.childrensoncologygroup.org/index.php/cog-family-handbook">https://www.childrensoncologygroup.org/index.php/cog-family-handbook</a>.

Visit the NCI's Web site at http://www.cancer.gov.





If you are in the United States, you may call the NCI's *Cancer Information Service* at: 1-800-4-CANCER (1-800-422-6237).

Information about long term follow-up after cancer treatment can be found at: http://www.survivorshipguidelines.org/.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You will get a copy of this form. You may also ask for a copy of the protocol (full study plan).

# Specimens for optional research tests

The choice to let us use specimens for research is up to you. No matter what you decide to do, it will not affect your care. You can still be a part of the main study even if you say 'No' to taking part in any of these optional research studies.

If you decide that your specimens can be used for research, some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

If you decide now that your specimens can be used for research, you can change your mind at any time. Just contact us and let us know that you do not want us to use your specimens. Then, any specimens that we have will be destroyed.

If you want to learn more about tissue research with specimens, the NCI website has an information sheet called "Providing Your Tissue For Research: What You Need To Know." This sheet can be found at: http://www.cancer.gov/clinicaltrials/resources/providingtissue.

Please read the information below and think about your choices. After making your decisions, check "Yes" or "No", then add your initials and the date after your answer. If you have any questions, please talk to your doctor or nurse, or call our research review board at the IRB's phone number included in this consent.

| 1.) | Please indicate by initialing below whether you choose to participate in the residual leukemia identification study. |
|---|---|
| | Yes No/ |
| 2.) | Please indicate by initialing below whether you choose to participate in the leukemid<br>immune cell ratio study. |
| | Yes No/ |





| 3.) | Please indicate by initialing below whether you choose to participate in the immune system study. | | | | | |
|---|---|---|---|---|---|---|
| | | Yes | . No | Initials | /<br>Date | |
| 4.) | Please indica<br>marker study. | | ng below whetl | ner you choose | to participate | e in the biological |
| | | Yes | . No | Initials | /<br>Date | |
| 5.) | Please indicate by initialing below whether you choose to participate in the flotetuze target quantification comparison study. | | | | | |
| | | Yes | . No | Initials | /<br>Date | |
| Sign | ature | | | | | |
| | e been given a<br>nment. | copy of al | l pages | of this form. T | he form inc | ludes one (1) |
| | reviewed the in<br>e to take part in | | | my questions an | swered. | |
| Partic | ipant | | | | | _Date |
| Paren | t/Guardian | | | | | _Date |
| Paren | t/Guardian | | | | | _Date |
| Physic | cian/PNP obtair | ning conser | nt | | | _Date |





## **Attachment 1**

## **Certificate of Confidentiality**

This trial is covered by a Certificate of Confidentiality from the federal government, which will help us protect the privacy of our research subjects. The Certificate protects against the involuntary release of information about subjects collected during the course of our covered studies. The researchers involved in the studies cannot be forced to disclose the identity or any information collected in the study in any legal proceedings at the federal, state, or local level, regardless of whether they are criminal, administrative, or legislative proceedings. However, the subject or the researcher may choose to voluntarily disclose the protected information under certain circumstances. For example, if the subject or his/her guardian requests the release of information in writing, the Certificate does not protect against that voluntary disclosure. Furthermore, federal agencies may review our records under limited circumstances, such as a DHHS request for information for an audit or program evaluation or an FDA request under the Food, Drug and Cosmetics Act. The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.